CLINICAL TRIAL: NCT01336049
Title: Nimotuzumab Plus Paclitaxel and Cisplatin as 1st Line Treatment for Esophageal Squamous Cell Cancer : a Single Center Prospective Clinical Trial
Brief Title: Nimotuzumab Plus Paclitaxel and Cisplatin as 1st Line Treatment for Esophageal Squamous Cell Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: zhang xiaodong, Peking University, School of Oncology, Department of GI oncology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N+TP-AEC3
Record Dates: First submitted 2011-03-29; First posted 2011-04-15 (Estimated); Last update posted 2011-04-15 (Estimated); Status verified 2011-03

CONDITIONS: Esophageal Squamous Cell Cancer
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — nimotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nimotuzumab (Experimental)
  Interventions: Drug: Nimotuzumab

INTERVENTIONS:
Drug: Nimotuzumab — Nimotuzumab 200mg/week

SUMMARY:
Nimotuzumab, as one new agent used in advanced esophageal carcinoma, has been shown to be effective and safe in some studies with head-neck cancers. Advanced esophageal carcinoma have poor prognosis and majority of patients resistant to chemotherapy in China. In the investigators phase II clinical trial proceeded before,the combination of paclitaxel with cisplatin showed good tolerance and efficacy to esophageal carcinoma. The investigators then initiated a prospective phase II clinical trial with Nimotuzumabplus paclitaxel/cisplatin as the 1st line treatment in advanced esophageal carcinoma to observe the efficacy and safety of the combination.

ELIGIBILITY:
Inclusion Criteria:

* Having signed informed consent
* Age 18 to 75 years old
* Histologically confirmed esophageal squamous carcinoma, Unresectable recurrent or metastatic disease,no prior palliative chemotherapy; No prior radiotherapy except radiotherapy at non-target lesion of the study more than 3 months,recurrence from last adjuvant chemotherapy or adjuvant radiotherapy should be longer than 6 months; no prior treatment of paclitaxel as adjuvant chemotherapy, total dose of cisplatin is less than 300mg/m2 if used in adjuvant chemotherapy
* Sex is not limited
* Measurable disease according to the RECIST criteria(diameter of the lesion should be more than 10mm by spiral CT or MRI, more than 20mm by common CT, the date of image should be less than 15 days before enrollment)
* Karnofsky performance status ≥80
* Life expectancy of ≥ 3 month
* WBC > 4,000/mm3, absolute neutrophil count ≥2000/mm3, platelet > 100,000/mm3, Hb > 10g/dl(within 14 days before enrollment),ALT and AST < 2.5 times ULN (≤5 times ULN in patients with liver metastases),Bilirubin level < 1.0 times ULN,Serum AKP < 2.5 times ULN,Serum creatinine < 1.0 times ULN
* No sever complication, such as active gastrointestinal bleeding, perforation, jaundice, obstruction, non-cancerous fever > 38℃；
* Normal ECG and heart function
* Fertile patients must use effective contraception
* Good compliance

Exclusion Criteria:

* Previous treatment of palliative chemotherapy or recurrence less than 6 months from time of last adjuvant chemo-/radiotherapy
* Known hypersensitivity to Nimotuzumab,Paclitaxel,Cisplatin
* Only with Brain or bone metastasis
* Tumor with length ≥ 10cm, liver metastasis covers more than 50% of liver,or lung metastasis covers more than 25% of lung
* No measurable lesions, eg. pleural fluid and ascites
* Suffer from severe heart disease or disease with other important organs
* Chronic diarrhea or renal dysfunction
* Pregnancy or lactation period
* Other previous malignancy within 5 year, except non-melanoma skin cancer
* Chronic diarrhea
* Mentally abnormal or disable cognition,including CNS metastasis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 6 weeks
  CT/MRI will be performed every 2 cycles of treatment for efficacy evaluation

SECONDARY OUTCOMES:
overall survival of all participants | 2 years
  OS means that from the first dose of treatment drug to death or lost, the follow-up visit will be performed every 3 months till death or lost
progression free survival | 1 year
  the follow-up visit of PFS will be performed every 2 cycles
adverse events | participants will be followed for the duration of hospital stay, an expected average of 1 week
  any adverse event will be record on CRF for safety control

CONTACTS AND LOCATIONS:
Locations (1):
- Xiaodong Zhang, Beijing, Beijing Municipality, China